CLINICAL TRIAL: NCT06866418
Title: Phagenyx® Registry Study: Evaluating Swallowing Therapy Outcomes and Recovery in the U.S.
Brief Title: Phagenyx® Registry Study
Acronym: RESTORE-US
Status: Recruiting | Type: Observational
Sponsor: Phagenesis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AHE-07
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control Group: Patient requires a nasogastric feeding tube for severe dysphagia and required dysphagia treatment
- Treatment Group: Patients who have undergone PES treatment for severe dysphagia.
  Interventions: Device: 1. Phagenyx® System Group Patients

INTERVENTIONS:
Device: 1. Phagenyx® System Group Patients — Patients who have undergone Pharyngeal Electrical Stimulation (PES) treatment for severe dysphagia using the Phagenyx® System
  Groups: Treatment Group

SUMMARY:
A retrospective, open-label, matched-control registry study designed to characterize the effectiveness of Pharyngeal Electrical Stimulation (PES) to improve swallowing in patients with severe dysphagia post stroke when delivered using the Phagenyx® System in real-world clinical settings in hospitals in the United States of America (US).

DETAILED DESCRIPTION:
The study will consist of a Treatment Group and a Control Group. The Treatment Group will include patients who have undergone PES treatment for severe dysphagia. The Control Group will consist of patients that qualify for PES treatment but are not treated with PES in the time period prior to implementing PES. Patients will be treated per standard of care at each institution. Each Treatment patient will receive treatment with PES in addition to other standard of care dysphagia therapies. Control subjects will receive standard of care dysphagia therapies only (no PES or other electrical stimulation therapies for dysphagia are permitted). Performance of the Phagenyx® System will be analyzed by comparing treatment outcomes for patients in the PES Group compared to patients in the Control Group.

The study will include patients with severe dysphagia post stroke. The main clinical outcomes will be assessed using the participating sites' standard of care methodology and will evaluate improvements in swallowing and reduction in associated treatments and complications.

ELIGIBILITY:
Inclusion Criteria:

1. Phagenyx® System Group Patients: Patients underwent treatment with the Phagenyx® System for a minimum of 3 treatments.
2. Control Group Patients: Patient requires a nasogastric feeding tube for severe dysphagia and required dysphagia treatment.
3. Willing and able to provide appropriate informed consent (if required).

Exclusion Criteria:

1. Primary endpoint outcome data not collected or not available.
2. In the investigator or sponsor's opinion the patient is not considered suitable.
3. Participation in another interventional study (medicinal or device) that could influence the outcomes of PES.
4. Treatment of dysphagia with other forms of electrical stimulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 600 patients total, comprised of 300 evaluable adult patients with severe dysphagia post stroke will be treated with PES with an additional 300 subjects enrolled as historical controls.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2036-09 (Estimated)

PRIMARY OUTCOMES:
Swallowing safety | Baseline to 2 (+1 days) post final PES treatment (Approximately 6 days).
  Swallowing safety based on the change in Penetration Aspiration Scale (PAS) score from baseline (pre-PES treatment) to 2 (+1 days) post PES treatment.
Nutritional Management | Baseline to Hospital Discharge (up to approximately 30 days)
  Nutritional management improvement based on the change in Functional Oral Intake Score (FOIS) from baseline (pre-PES treatment) to hospital discharge

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - HMH Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No